CLINICAL TRIAL: NCT00270621
Title: Family Help Program: Primary Care Delivery by Telephone for Psychological and Behavioural Problems (Pediatric Enuresis)
Brief Title: Family Help Program: Nighttime Enuresis Treatment Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2234e; CIHR CAHR-43273 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Enuresis
MeSH Terms: conditions — Enuresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): FHP Night time Enuresis intervention
  Interventions: Behavioral: FHP Night time ENuresis Intervention
- Control (No Intervention): To receive standard/usual care for Nocturnal Enuresis- No FHP Night time Enuresis INtervention

INTERVENTIONS:
Behavioral: FHP Night time ENuresis Intervention — Urine alarm/evidence-based psychological Intervention
  Arms: Treatment

SUMMARY:
The purpose of the Strongest Families (formerly Family Help Program)is to evaluate the effectiveness of the Strongest Families distance intervention compared to usual or standard care that is typically provided to children with mild to moderate Enuresis diagnoses. This is a single-centre trial based at the IWK Health Centre. The primary outcome is change in diagnosis.

DETAILED DESCRIPTION:
The purpose of the Family Help Program is to deliver, primary care mental health services to children and their families in the comfort and privacy of their own home. Approximately 46 children (5-12 years of age)suffering from pediatric enuresis (at least 2 times a week) will be randomized.

The intervention is delivered from a distance, using the urine alarm system accompanied by educational materials (manuals, video-tapes, audio-tapes) and telephone consultation with a trained paraprofessional "coach" who is supervised by a licensed health care professional. The telephone coach delivers consistent care based on written protocols, with on-going evaluation by a professional team.

Fifty percent of the eligible participants will receive Family Help Program telephone-based treatment and 50% will be referred back to their family physician to receive standard care as determined by that physician. Those receiving standard care will be evaluated for outcome results and then compared to the Family Help treated participants. It is anticipated that Family Help treatment will be proven to be as or more effective than standard care.

ELIGIBILITY:
Inclusion Criteria:

* Is your child 3 to 12 years of age
* child wets the bed more than twice per week
* child dry during the day

Exclusion Criteria:

* child received any treatment for bedwetting in the past 6 months
* child at any time been dry for 6 months or longer
* child currently on Imipramine or Desmopressin

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Diagnosis using KSADS at baseline, 120, 240 and 365 day follow-up. | baseline, 120, 240 and 365 day follow-up

SECONDARY OUTCOMES:
Symptomology frequency as evidenced by diary data; | daily during treatment; 3 weeks on follow-up at 240 & 365 day post randomization
Disability Measure; | weekly during treatment; baseline, 120, 240 and 365 day follow-up
Child Health Questionnaire | baseline, 120, 240 and 365 day follow-up
Economic Outcome assessment | baseline, 120, 240 and 365 day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. McGrath, PhD., Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate summary data would be made available but not individual data.

REFERENCES:
- [Background] Lingley-Pottie P, McGrath PJ. A paediatric therapeutic alliance occurs with distance intervention. J Telemed Telecare. 2008;14(5):236-40. doi: 10.1258/jtt.2008.080101. PMID 18632997
- [Background] Lingley-Pottie P, McGrath PJ. Telehealth: a child and family-friendly approach to mental health-care reform. J Telemed Telecare. 2008;14(5):225-6. doi: 10.1258/jtt.2008.008001. PMID 18632994
- [Background] McGrath PJ, Lingley-Pottie P, Emberly DJ, Thurston C, McLean C. Integrated knowledge translation in mental health: family help as an example. J Can Acad Child Adolesc Psychiatry. 2009 Feb;18(1):30-7. PMID 19270846
- [Result] Lingely-Pottie P, McGrath PJ. A therapeutic alliance can exist without face-to-face contact. J Telemed Telecare. 2006;12(8):396-9. doi: 10.1258/135763306779378690. PMID 17227604
- [Result] Lingley-Pottie P, McGrath PJ. Distance therapeutic alliance: the participant's experience. ANS Adv Nurs Sci. 2007 Oct-Dec;30(4):353-66. doi: 10.1097/01.ANS.0000300184.94595.25. PMID 18025870
- [Derived] Caldwell PH, Codarini M, Stewart F, Hahn D, Sureshkumar P. Alarm interventions for nocturnal enuresis in children. Cochrane Database Syst Rev. 2020 May 4;5(5):CD002911. doi: 10.1002/14651858.CD002911.pub3. PMID 32364251
- See also: Family Help Program — http://www.bringinghealthhome.com/